CLINICAL TRIAL: NCT01594476
Title: Early Versus Standard Interval Postpartum Intrauterine Device (IUD) Placement at 3 Weeks or 6 Weeks Following Delivery: A Prospective Randomized Trial
Brief Title: Early Postpartum Intrauterine Device (IUD) Placement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Incomplete study enrollment prior to depletion of funding
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Maureen Baldwin, Instructor, Ob/Gyn, Fellow in Family Planning, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8120
Record Dates: First submitted 2012-03-09; First posted 2012-05-09 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Contraception
Keywords: Postpartum; Contraception; Intrauterine device; Intrauterine system; Mirena; Paragard; Uterine involution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levonorgestrel IUS insertion at 3 weeks (Experimental): IUD placement at 3 weeks after delivery.
  Interventions: Drug: Levonorgestrel IUS
- Levonorgestrel IUS insertion at 6 weeks (Experimental): IUD placement at 6 weeks after delivery.
  Interventions: Drug: Levonorgestrel IUS

INTERVENTIONS:
Drug: Levonorgestrel IUS — 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
  Other Names: Mirena IUS; Paragard IUD

SUMMARY:
Women who have just given birth are at high risk for rapid repeat pregnancy, which can lead to negative consequences during the subsequent pregnancy. Providers have traditionally delayed starting birth control, especially placement of intrauterine devices (IUDs), post-delivery for a number of reasons. The first postpartum visit after a woman has given birth is typically scheduled for 6 weeks after her delivery, during which she is typically provided with her chosen method of birth control. This study will evaluate two different IUD placement times: 3 weeks and 6 weeks after delivery. This will allow the researchers to determine if placement time affects a woman's follow-through obtaining the IUD and keeping it inserted in place. The researchers will also look at bleeding patterns and patient/provider satisfaction with the IUD placement

DETAILED DESCRIPTION:
The goal of this study is to investigate whether early interval placement of a postpartum IUD at 3 weeks postpartum, compared to the usual 6 weeks postpartum, is associated with greater uptake of the IUD by 3 months after delivery. Many women do not return for a follow up visit. We will investigate whether they are more likely to return and to receive an IUD if the follow up visit is earlier. Measures of 6 month IUD continuation, subject acceptability, safety and efficacy will also be examined. This prospective, randomized, controlled trial will enroll approximately 240 women at our academic tertiary care hospital in the United States. Participants will be recruited from women who deliver a live-born singleton infant at greater than 32 weeks gestation and who have indicated interest in obtaining intrauterine contraception. Subjects will choose to receive either a levonorgestrel-containing IUS (Mirena) or copper T380A IUD (ParaGard). Enrolled subjects will be randomized to IUD placement at either 3 weeks (+/- 3 days) or 6 weeks (+/- 3 days) after their delivery date. Women will be followed by phone contacts at 3 months and 4 months and will have a clinic visit with an ultrasound at 6 months after delivery. The IUD position in the uterus and the uterine size will be assessed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* Voluntarily requesting either copper T380A or levonorgestrel IUD placement for postpartum contraception
* Within 5 days of vaginal or cesarean delivery of live born infant ≥32 0/7 weeks at the time of enrollment
* English or Spanish speaking
* Able to give consent and agree to terms of the study
* No contraindications to use of either intrauterine device

Exclusion Criteria:

* Preterm delivery prior to 32 weeks gestation
* Recent pregnancy with multiple gestation
* Current incarceration
* Known congenital or acquired uterine anomaly, including fibroids that distort the uterine cavity
* Current or recent pelvic infection (chorioamnionitis treated for fever in labor only is not an exclusion)
* Suspected hypersensitivity or contraindication to the chosen IUD
* No insurance coverage for postpartum care, including Citizen Alien Waived Emergent Medical (CAWEM)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Baldwin, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Baldwin MK, Hart KD, Rodriguez MI. Predictors for follow-up among postpartum patients enrolled in a clinical trial. Contraception. 2018 Sep;98(3):228-231. doi: 10.1016/j.contraception.2018.04.016. Epub 2018 May 8. PMID 29750924

RESULTS

PARTICIPANT FLOW:
Groups:
- IUD Insertion at 3 Weeks: IUD placement at 3 weeks after delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS or Copper T intrauterine device
- IUD Insertion at 6 Weeks: IUD placement at 6 weeks after delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS or Copper T intrauterine device
Period: Overall Study
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Started | 101 | 100
Received Intervention | 66 | 73
Excluded After Allocation | 1 | 3
IUD Removal (By 6 months) | 3 | 5
IUD Expulsion (By 6 months) | 2 | 0
Pregnant (By 6 months None had IUD in place at the time of pregnancy) | 2 | 5
Completed (Analyzed for intent to treat) | 100 | 97
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levonorgestrel IUS Insertion at 3 Weeks | Levonorgestrel IUS Insertion at 6 Weeks | Total
Number analyzed (Participants) | 100 | 97 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (5.7) | 29.0 (5.8) | 28.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 97 | 197
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 86 | 84 | 170
  Unknown or Not Reported | 0 | 0 | 0
Insurance type [Count of Participants; unit: Participants]
  Public insurance | 48 | 47 | 95
  Private insurance | 52 | 50 | 102
Planned pregnancy [Count of Participants; unit: Participants]
  Unplanned | 49 | 48 | 97
  Planned | 51 | 49 | 100
Delivery type [Count of Participants; unit: Participants]
  Vaginal | 75 | 71 | 146
  Cesarean | 25 | 26 | 51
Education [Count of Participants; unit: Participants]
  High school/GED or less | 31 | 23 | 54
  More than high school | 69 | 74 | 143
Snyder Hope Scale [Mean (Standard Deviation); unit: units on a scale] — The Snyder Hope Scale (Future Scale) is a 12-question validated survey that includes four questions that reflect agency, four that reflect pathways, and four that are distracters. Responses to this scale correlate well with other psychological tests designed to assess optimism, expectancy for attaining goals, and self-esteem. The distracter questions are not scored. The maximum total score is 64 (range 0-64; max 8 points per 8 questions scored and added). Each subscale has a maximum total score of 32 (range 0-32). Higher total score and subscale scores indicate better agency and pathways.
  units on a scale
    Future Scale total score | 47.2 (5.4) | 45.9 (6.7) | 46.5 (6.1)
    Agency subscale score | 23.8 (3.0) | 22.9 (4.1) | 23.4 (3.6)
    Pathway subscale score | 23.4 (3.2) | 22.8 (3.8) | 23.1 (3.5)
Social-Support Scale [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Scale of Perceived Social Support (MDSS) is a 12-question validated survey to assess perceived social support, another possible indicator for the ability to carry out a plan. The scores can be separated into 3 subscale domains for perceived support from family, friends, and significant other. Maximum total score is 84 (range 0-84), which included added subscale scores of maximum 28 (0-28) for 4 questions each. Higher scores indicate more perceived social support.
  units on a scale
    MDSS total score | 65.8 (9.0) | 63.5 (10.7) | 64.7 (9.8)
    Family subscale score | 22.0 (3.6) | 20.4 (5.6) | 21.2 (4.7)
    Friends subscale score | 21.3 (4.2) | 20.5 (5.2) | 20.9 (4.7)
    Significant other subscale score | 23.0 (2.0) | 22.4 (3.2) | 22.7 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With an IUD at 3 Months Postpartum
Description: Subjects will be contacted by phone or email at 3 months after delivery. We will compare the proportion of subjects who report having an IUD in place at 3 months after delivery of those who are randomized to each group (placement at either 3 weeks or 6 weeks) .
Time Frame: Three months after delivery
Population: Data analyzed as intent to treat regardless of when they had their IUD placed. This is IUD placed by 3 months in each group.
Measure: Count of Participants; unit: Participants
Groups:
- IUD Insertion at 3 Weeks: IUD placement at 3 weeks after delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
- IUD Insertion at 6 Weeks: IUD placement at 6 weeks after delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Number analyzed (Participants) | 100 | 97
Participants | 66 | 73

2. Secondary Outcome: Satisfaction With the Timing of IUD Placement.
Description: Subjects were asked to record their overall satisfaction with the timing of the IUD placement on a 100 millimeter (mm) visual analog scale (VAS). A VAS is a 100 mm horizontal line with anchors stating "very dissatisfied" and "very satisfied." The VAS score is calculated by measuring the distance in millimeters between the left end of the scale and the intersection of a vertical mark placed by the subject. Maximum score is 100 (range 0-100). Higher scores indicate higher satisfaction.
Time Frame: Immediately following IUD placement.
Population: Includes all subjects enrolled on protocol who underwent IUD placement at a study visit at any timing prior to 3 months postpartum. Comparison is based on randomization timing but actual timing of placement may have differed. Numbers differ from primary outcome due to removals and expulsion prior to 3 months, and placement outside study visits.
Measure: Mean (Standard Deviation); unit: mm on VAS
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Number analyzed (Participants) | 68 | 68
mm on VAS | 90.6 (17.2) | 93.5 (12.0)

3. Secondary Outcome: Uterine Thickness at the Fundus
Description: Transvaginal ultrasound will be performed immediately following IUD placement. The thickness of the uterine myometrium at the fundus from the endometrium to the outer edge of the serosa will be measured in centimeters using an ultrasound caliper in the sagittal view.
Time Frame: At IUD placement
Population: Subjects who had their IUD placed at the allocated timing of 18-24 days versus 39-45 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Number analyzed (Participants) | 54 | 61
cm | 2.3 (0.8) | 1.7 (0.4)

4. Secondary Outcome: Subjects With an IUD at 6 Months Postpartum
Description: Subjects will return to clinic for an ultrasound and exam at six months after delivery. We will compare the proportion of subjects with an IUD at this time of those randomized to each placement timing.
Time Frame: Six months after delivery
Population: Population is subject randomization groups.
Measure: Count of Participants; unit: Participants
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Number analyzed (Participants) | 100 | 97
Participants | 53 | 53

5. Secondary Outcome: Number of Subjects With Adverse Events
Description: Subjects will be followed for 6 months each. Over the 6 month study period, the number and proportion of subjects who experience adverse events including treatment for infection, IUD expulsion or IUD perforation will be assessed.
Time Frame: Six months after delivery
Population: All subjects analyzed. This includes all subjects enrolled on protocol and allocated. There were no adverse events in the subjects excluded after allocation.
Measure: Count of Participants; unit: Participants
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Number analyzed (Participants) | 100 | 97
Participants
  IUD expulsion | 2 | 0
  IUD perforation | 0 | 0
  Pregnancy with IUD in place | 0 | 0
  Infection with IUD in place | 0 | 0
  No known adverse events | 98 | 97

6. Secondary Outcome: Pain With IUD Placement
Description: Subjects were asked to record their current pain immediate at the time of the IUD placement on a 100 millimeter (mm) visual analog scale (VAS). A VAS is a 100 mm horizontal line with anchors stating "no pain" and "worst pain in my life." The VAS score is calculated by measuring the distance in millimeters between the left end of the scale and the intersection of a vertical mark placed by the subject. Maximum score is 100 (range 0-100). Higher scores indicate higher pain. The distance from the left side of the 10 cm line to the mark will be measured in millimeters and compared between randomization groups if they received an IUD at the allocated timing of 18-24 or 39-45 days.
Time Frame: At the time of IUD placement.
Population: Subjects analyzed by actual timing of IUD insertion
Measure: Mean (Standard Deviation); unit: mm
Groups:
- 18-24 Days After Vaginal Delivery: IUD placement at 18-24 days after vaginal delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
- 39-45 Days After Vaginal Delivery: IUD placement at 39-45 days after vaginal delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
- 18-24 Days After Cesarean Delivery: IUD placement at 18-24 days after cesarean delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
- 39-45 Days After Cesarean Delivery: IUD placement at 39-45 days after cesarean delivery.
  Levonorgestrel IUS: 20 mcg levonorgestrel per day in intrauterine system for Mirena IUS Copper T intrauterine device
Arm/Group | 18-24 Days After Vaginal Delivery | 39-45 Days After Vaginal Delivery | 18-24 Days After Cesarean Delivery | 39-45 Days After Cesarean Delivery
Number analyzed (Participants) | 39 | 47 | 16 | 14
mm | 15.7 (16.4) | 23.0 (21.0) | 30.9 (27.3) | 32.1 (27.9)

ADVERSE EVENTS:
Arm/Group | IUD Insertion at 3 Weeks | IUD Insertion at 6 Weeks
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/97
Other Adverse Events (participants affected / at risk) | 2/100 | 0/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IUD Insertion at 3 Weeks (N=100) | IUD Insertion at 6 Weeks (N=97)
IUD expulsion (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Partial or complete expulsion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No